CLINICAL TRIAL: NCT03092960
Title: The HOMBRE Trial: Comparing Two Innovative Approaches to Reduce Chronic Disease Risk Among Latino Men
Acronym: HOMBRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Medical Foundation (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Illinois at Chicago (Other); RTI International (Other); University of Pittsburgh (Other); Arizona State University (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 981746
Record Dates: First submitted 2017-03-15; First posted 2017-03-28 (Actual); Results first posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Obesity; Metabolic Syndrome; Lifestyle Intervention; Pre Diabetes
Keywords: Latino; Male
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Glucose Intolerance

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal intensity intervention (Active Comparator): Patients assigned to this group will received the Minimal intensity intervention.
  Interventions: Behavioral: Minimal intensity intervention
- HOMBRE (Experimental): Patients assigned to this group will receive the HOMBRE intervention
  Interventions: Behavioral: HOMBRE

INTERVENTIONS:
Behavioral: Minimal intensity intervention — The minimal intensity intervention control includes the Group Lifestyle Balance (GLB) videos (DVD or online), standardized messages, and access to a lifestyle coach if initiated by the participant.
  Arms: Minimal intensity intervention
Behavioral: HOMBRE — HOMBRE is a Group Lifestyle Balance (GLB)-based intervention tailored for men and available in 3 delivery modalities (coach-facilitated individual approach, coach-led online virtual groups, and coach-led in-person groups). A lifestyle coach will support men in making an informed choice of modality and will provide ongoing individualized feedback. All delivery modalities provide the same evidence-based curriculum and include self-monitoring and individualized feedback from the lifestyle coach.
  Arms: HOMBRE

SUMMARY:
The purpose of this study is to test a flexible lifestyle program designed to help Latino men make healthy lifestyle changes to lower their risk of developing diabetes and heart disease. The program is called HOMBRE (Hombres con Opciones para Mejorar el Bienestar y bajar el Riesgo de Enfermedades crónicas; English translation: Men with choices to improve well being and decrease chronic disease risk).

DETAILED DESCRIPTION:
This study is a comparative effectiveness trial where obese Latino men will receive, by random assignment, the HOMBRE intervention or a minimal intensity intervention.

The study is designed to test whether a flexible lifestyle program with choices for program engagement will lead to better health outcomes, compared to a minimal intensity self-directed lifestyle program. If proven successful, this study has the potential to significantly impact health outcomes that matter to Latino men through the innovative design of lifestyle interventions to prevent chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* Latino of any race
* BMI >27 kg/m2
* One or more metabolic syndrome component (high triglycerides, blood pressure, fasting glucose, central obesity, or low HDL cholesterol)
* Primary Care Physician approval of patient study contact
* Able and willing to enroll and provide informed consent, i.e., to meet the time and data collection requirements of the study, be randomized to one of tow study arms, participate in follow-up for 18 months, and authorize the extraction of relevant information form the Electronic Health Record.

Exclusion Criteria:

Medical exclusions:

* Previous diagnosis of diabetes or diabetes diagnosed as a result of fasting blood glucose or hemoglobin A1c levels obtained through study screening;
* Diagnosis of cancer (other than non-melanoma skin cancer) that is/was active or treated with radiation or chemotherapy within the past 2 years;
* Inability to walk without the assistance of another person;
* Severe medical co-morbidities that require aggressive treatment: e.g., stage 4 or greater renal disease, class III or greater heart failure, unstable coronary artery disease, liver or renal failure;
* Diagnosis of a terminal illness and/or in hospice care;
* Diagnosis of bipolar disorder or psychotic disorder within the last 2 years, or currently taking a mood stabilizer or antipsychotic medication
* Initiation or change in type or dosing of antidepressant medications within 2 months prior to enrollment (The patient will be re-contacted for a later cohort once his/her regimen has been stable for at least 2 months unless the person declines to participate altogether.)
* Have had or plan to undergo bariatric surgery during the study period

Other exclusions:

* Having no reliable telephone service
* Plan to move out of the area during the study period
* Family/household member of another study participant or of a study staff member
* Investigator discretion for clinical safety or protocol adherence reasons

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identifies as male.
Enrollment: 424 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Goldman Rosas, PhD, MPH, Principal Investigator — Stanford University; Kristen M Azar, RN, MSN, MPH, Principal Investigator — Sutter Health Research Development & Dissemination
Locations (1):
- Palo Alto Medical Foundation, Palo Alto, California, United States

REFERENCES:
- [Derived] Rosas LG, Lv N, Xiao L, Venditti EM, Lewis MA, Azar KMJ, Hooker SP, Zavella P, Ma J. HOMBRE: A Trial Comparing 2 Weight Loss Approaches for Latino Men. Am J Prev Med. 2022 Sep;63(3):341-353. doi: 10.1016/j.amepre.2022.03.032. Epub 2022 May 30. PMID 35654660
- [Derived] Rosas LG, Lv N, Xiao L, Azar KM, Hooker SP, Venditti EM, Lewis MA, Zavella P, Ma J. Preferences for Technology-Mediated Behavioral Lifestyle Interventions With Different Levels of Coach and Peer Support Among Latino Men: Comparative Study Within One Arm of a Randomized Controlled Trial. JMIR Form Res. 2022 Feb 4;6(2):e29537. doi: 10.2196/29537. PMID 35119377

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Minimal Intensity Intervention | HOMBRE
Started | 212 | 212
Completed | 180 | 186
Not Completed | 32 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minimal Intensity Intervention | HOMBRE | Total
Number analyzed (Participants) | 212 | 212 | 424
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (12.1) | 47.0 (11.8) | 47.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 212 | 212 | 424
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 212 | 212 | 424
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 212 | 212 | 424
Weight, kg [Mean (Standard Deviation); unit: kg] | 99.2 (17.9) | 101.5 (33.0) | 100.4 (26.6)

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Men Achieving 5% Weight Loss or More
Description: Number and Percentage of men who achieve 5% or more of weight loss compared to their baseline weight
Time Frame: Baseline, 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 180 | 186
Participants | 37 | 51

2. Secondary Outcome: Trajectory of Weight Change From Baseline Through 18 Months
Description: Slope of changes in weights abstracted from EHR from baseline through 18 months
Time Frame: 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. For examining weight loss trajectory over time, we abstracted weight measurements from the EHR from 3 months prior to randomization to 24 months post randomization. 209 in HOMBRE and 209 in Minimal Intensity intervention had EHR-abstracted weight during this 27-month period.
Measure: Mean (Standard Deviation); unit: kg/month
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 209 | 209
kg/month | -0.11 (0.04) | -0.13 (0.04)

3. Secondary Outcome: Changes in Weight From Baseline
Description: Weight measurements were abstracted from EHR.
Time Frame: 6 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. We used same model as first secondary outcome to examine changes in EHR weight at 6 months. We abstracted weight from the EHR from 3 months prior to randomization to 24 months post randomization. 209 in HOMBRE and 209 in Minimal Intensity had EHR-abstracted weight during this 27-month period.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 209 | 209
kg | -1.79 (6.10) | -2.78 (5.45)

4. Secondary Outcome: Changes in Weight From Baseline
Description: Weight measurements were abstracted from EHR.
Time Frame: 12 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity had either study-measured, EHR-abstracted, or self-reported weight, therefore were counted in retention in the Participant Flow module. We used same model as first secondary outcome to examine changes in EHR weight at 12 months. We abstracted weight from the EHR from 3 months prior to randomization to 24 months post randomization. 209 in HOMBRE and 209 in Minimal Intensity had EHR-abstracted weight during this 27-month period.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 209 | 209
kg | -1.56 (7.00) | -2.77 (6.47)

5. Secondary Outcome: Changes in Weight From Baseline
Description: Weight measurements were abstracted from EHR.
Time Frame: 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity had either study-measured, EHR-abstracted, or self-reported weight, therefore were counted in retention in the Participant Flow module. We used same model as first secondary outcome to examine changes in EHR weight at 18 months. We abstracted weight from the EHR from 3 months prior to randomization to 24 months post randomization. 209 in HOMBRE and 209 in Minimal Intensity had EHR-abstracted weight during this 27-month period.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 209 | 209
kg | -1.67 (6.16) | -2.46 (6.60)

6. Secondary Outcome: Change in Waist Circumference From Baseline
Description: Waist circumference at 18 months - waist circumference at baseline
Time Frame: Baseline, 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. Among them 83 in the HOMBRE intervention and 88 in the Minimal Intensity intervention had waist circumference data at 18 months.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 88 | 83
cm | -0.0 (6.7) | -0.8 (5.7)

7. Secondary Outcome: Change in Systolic Blood Pressure From Baseline
Description: Systolic blood pressure at 18 months - systolic blood pressure at baseline
Time Frame: Baseline, 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. Among them 147 in the HOMBRE intervention and 145 in the Minimal Intensity intervention had blood pressure data at 18 months.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 145 | 147
mm Hg | 0.4 (12.5) | 0.8 (11.6)

8. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline
Description: Diastolic blood pressure at 18 months - diastolic blood pressure at baseline
Time Frame: Baseline, 18 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 145 | 147
mm Hg | -2.7 (9.4) | -2.3 (9.0)

9. Secondary Outcome: Change in Health Behavior: Leisure Time Physical Activity
Description: Physical activity measured at 18 months minus physical activity measured at baseline using Stanford 7-day physical activity recall
Time Frame: Baseline, 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. Among them 174 in the HOMBRE intervention and 177 in the Minimal Intensity intervention had physical activity data at 18 months.
Measure: Mean (Standard Deviation); unit: MET minutes/week
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 177 | 174
MET minutes/week | -113 (1410) | -369 (1436)

10. Secondary Outcome: Change in Health Behavior: Energy Expenditure
Description: The Stanford 7-day Physical Activity Recall data also provided estimates of total daily energy expenditures. Total energy expenditure = sleep hours × 1 MET + light activity hours × 1.5 METs + moderate activity hours × 4 METs + hard activity hours × 6 METs + very hard activity hours × 10 METs. Total daily energy expenditure at 18 months - Total daily energy expenditure at baseline.
Time Frame: Baseline, 18 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: kcal/kg/day
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 177 | 174
kcal/kg/day | -1.1 (5.3) | -2.1 (6.0)

11. Secondary Outcome: Change in Health Behavior: Sedentary Behavior
Description: Weekly hours of sedentary behavior measured at 18 months minus weekly hours of sedentary behavior at baseline using the Sedentary behavior Questionnaire
Time Frame: Baseline, 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. Among them 136 in the HOMBRE intervention and 137 in the Minimal Intensity intervention had sedentary behavior data at 18 months.
Measure: Mean (Standard Deviation); unit: hours/week
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 137 | 136
hours/week | -1.5 (31.5) | -2.4 (47.5)

12. Secondary Outcome: Change in Health Behavior: Diet Quality
Description: Dietary intake was measured using the gold-standard approach of multiple pass 24-hour recalls in Spanish or English using Nutrition Data System for Research (NDSR). Diet quality was assessed by the Dietary Approaches to Stop Hypertension (DASH) score. DASH scores were calculated based on combining nine nutrient targets (i.e. total fat, saturated fat, protein, cholesterol, fiber, magnesium, calcium, sodium and potassium). A higher score reflects higher diet quality. The minimum score is 8 and the maximum is 40. DASH score at 18 months - DASH score at baseline.
Time Frame: Baseline, 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. Among them 80 in the HOMBRE intervention and 90 in the Minimal Intensity intervention had diet data at 18 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 90 | 80
score on a scale | 0.2 (1.9) | 0.3 (1.8)

13. Secondary Outcome: Change in Health Behavior: Fruit and Vegetable Intake
Description: Fruit and vegetable intake measured at 18 months minus fruit and vegetable intake measured at baseline using 24-hour multiple pass recalls. Fruit and vegetable intake is measured in servings per day.
Time Frame: Baseline, 18 months
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: servings/day
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 90 | 80
servings/day | 0.3 (4.1) | -0.4 (3.8)

14. Secondary Outcome: Change in Health Behavior: Total Calorie Intake
Description: Total calorie intake per day measured at 18 months minus total calorie intake per day measured at baseline using 24-hour multiple pass dietary recalls.
Time Frame: Baseline, 18 months
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: kilocalories/day
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 90 | 80
kilocalories/day | 4.0 (3.8) | 4.1 (3.0)

15. Secondary Outcome: Change in Health Behavior: Total Fat
Description: Total fat consumption per day measured at 18 months minus total fat consumption per day measured at baseline using 24-hour multiple pass dietary recalls.
Time Frame: Baseline, 18 months
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 90 | 80
g/day | -23.2 (121) | -14.8 (44.9)

16. Secondary Outcome: Change in Psychosocial Well-being: Obesity-specific Quality of Life
Description: Obesity-related Problem Scale, average scores of 8 questions with a range from 0 (no at all) to 3 (extremely). The average score is then multiplied by 100 and divided by 3 to convert to a scale of 0-100, with a higher score indicating more obesity-related problems. Obesity-related quality of life measured at 18 months - obesity-related quality of life measured at baseline.
Time Frame: Baseline, 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. Among them 105 in the HOMBRE intervention and 101 in the Minimal Intensity intervention had obesity-related quality of life data at 18 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 101 | 105
units on a scale | -6.3 (21.4) | -7.4 (19.9)

17. Secondary Outcome: Change in Psychosocial Well-being: Depressive Symptoms
Description: The Patient Health Questionnaire PHQ-9 is a self-report questionnaire with 9 items. Respondents answered questions regarding how often a symptom has bothered them over the last two weeks. Each item is rated on a 4-point scale (0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day). PHQ-9 total score is the sum of the nine items, ranging from 0 to 27. Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively. PHQ-9 score at 18 months - PHQ-9 score at baseline.
Time Frame: Baseline, 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. Among them 104 in the HOMBRE intervention and 101 in the Minimal Intensity intervention had depression symptom data at 18 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 101 | 104
score on a scale | -0.8 (3.9) | -0.6 (3.8)

18. Secondary Outcome: Change in Perceived Stress
Description: Perceived stress scale with a range of 0 to 40 with higher scores indicating higher stress. Perceived stress at 18 months - Perceived stress at baseline.
Time Frame: Baseline, 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. Among them 105 in the HOMBRE intervention and 101 in the Minimal Intensity intervention had perceived stress data at 18 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 101 | 105
score on a scale | 0.0 (5.6) | -1.1 (5.6)

19. Secondary Outcome: Change in Psychosocial Well-being: Sleep Disturbance T-score
Description: Sleep disturbance T-score, a population scale with a range from 25 (extreme disturbance or impairment) to 80 (not at all) converted from the raw total score of 8-item questionnaire. A score of 50 represents the average of the calibration sample, which was generally more enriched for chronic illness. Sleep disturbance score at 18 months - sleep disturbance score at baseline.
Time Frame: Baseline, 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. Among them 103 in the HOMBRE intervention and 100 in the Minimal Intensity intervention had sleep disturbance data at 18 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 100 | 103
score on a scale | -0.7 (8.2) | -0.2 (7.7)

20. Secondary Outcome: Change in Psychosocial Well-being: Sleep Impairment T-score
Description: Sleep Impairment T-score, a population scale with a range from 25 (extreme disturbance or impairment) to 80 (not at all) converted from the raw total score of 8-item questionnaire. A score of 50 represents the average of the calibration sample, which was generally more enriched for chronic illness. Sleep impairment score at 18 months - sleep impairment at baseline.
Time Frame: Baseline, 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. Among them 103 in the HOMBRE intervention and 100 in the Minimal Intensity intervention had sleep impairment data at 18 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 100 | 103
score on a scale | -0.1 (9.3) | -2.9 (9.2)

21. Secondary Outcome: Psychosocial Well-being: Number and Percentage of Participants Who Had no Problems With Mobility Domain in Utility-based Quality of Life Measured by EuroQol EQ-5D
Description: Utility-based quality of life was measured by EuroQol EQ-5D. Number and percentage of participants who had no problems with mobility.
Time Frame: 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. Among them 107 in the HOMBRE intervention and 104 in the Minimal Intensity intervention had utility-based quality of life mobility data at 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 104 | 107
Participants | 91 | 96

22. Secondary Outcome: Change in Psychosocial Well-being: Number and Percentage of Participants Who Had no Problems With Self Care Domain in Utility-based Quality of Life Measured by EuroQol EQ-5D
Description: Number and percentage of participants who had no problems with self care was measured using the Euro-QoL 5D (EQ-5D-5L), which includes 5 domains (mobility, self-care, usual activities, pain and discomfort, and depression and anxiety) scored on 5 levels (no, slight, moderate, severe, or extreme problems) and current health rated on a visual analogue scale from 0 to 100.
Time Frame: 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. Among them 108 in the HOMBRE intervention and 104 in the Minimal Intensity intervention had utility-based quality of life - self care data at 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 104 | 108
Participants | 101 | 106

23. Secondary Outcome: Change in Psychosocial Well-being: Number and Percentage of Participants Who Had no Problems With Usual Activities Domain in Utility-based Quality of Life Measured by EuroQol EQ-5D
Description: Number and percentage of participants who had no problems with usual activities (e.g. work, study, housework, family or leisure activities).
Time Frame: 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. Among them 108 in the HOMBRE intervention and 104 in the Minimal Intensity intervention had utility-based quality of life usual activity data at 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 104 | 108
Participants | 96 | 97

24. Secondary Outcome: Change in Psychosocial Well-being: Number and Percentage of Participants Who Had no Problems With Pain/Discomfort Domain in Utility-based Quality of Life Measured by EuroQol EQ-5D
Description: Number and percentage of participants who had no problems with pain was measured using the Euro-QoL 5D (EQ-5D-5L), which includes 5 domains (mobility, self-care, usual activities, pain and discomfort, and depression and anxiety) scored on 5 levels (no, slight, moderate, severe, or extreme problems) and current health rated on a visual analogue scale from 0 to 100.
Time Frame: 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. Among them 108 in the HOMBRE intervention and 104 in the Minimal Intensity intervention had utility-based quality of life pain/discomfort data at 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 104 | 108
Participants | 55 | 66

25. Secondary Outcome: Change in Psychosocial Well-being: Number and Percentage of Participants Who Had no Problems With Anxiety and Depression Domain in Utility-based Quality of Life Measured by EuroQol EQ-5D
Description: Number and percentage of participants who had no problems with anxiety and depression was measured using the Euro-QoL 5D (EQ-5D-5L), which includes 5 domains (mobility, self-care, usual activities, pain and discomfort, and depression and anxiety) scored on 5 levels (no, slight, moderate, severe, or extreme problems) and current health rated on a visual analogue scale from 0 to 100.
Time Frame: 18 months
Population: At 18 months, 186 in HOMBRE and 180 in Minimal Intensity intervention had either study-measured weight, EHR-abstracted weight, or self-reported weight, therefore were counted in retention in the Participant Flow module. Among them 108 in the HOMBRE intervention and 104 in the Minimal Intensity intervention had utility-based quality of life anxiety/depression data at 18 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Minimal Intensity Intervention | HOMBRE
Number analyzed (Participants) | 104 | 108
Participants | 72 | 85

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Minimal Intensity Intervention | HOMBRE
All-Cause Mortality (participants affected / at risk) | 0/212 | 0/212
Serious Adverse Events (participants affected / at risk) | 15/212 | 14/212
Other Adverse Events (participants affected / at risk) | 48/212 | 52/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minimal Intensity Intervention (N=212) | HOMBRE (N=212)
Endocrine disorders (Endocrine disorders) | 3 (3) | 0 (0)
Gastrointestinal Disorders (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immune System Disorders (Immune system disorders) | 0 (0) | 1 (2)
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (11)
Renal and Urinary Disorders (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Cardiac disorders (Cardiac disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minimal Intensity Intervention (N=212) | HOMBRE (N=212)
Endocrine Disorders (Endocrine disorders) | 1 (1) | 0 (0)
Gastrointestinal Disorders (Gastrointestinal disorders) | 1 (1) | 3 (3)
General disorders (General disorders) | 2 (2) | 6 (7)
Infections and Infestations (Infections and infestations) | 2 (4) | 0 (0)
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 34 (41) | 28 (35)
Nervous System Disorders (Nervous system disorders) | 2 (2) | 2 (2)
Renal and Urinary Disorder (Renal and urinary disorders) | 2 (2) | 0 (0)
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Cardiac disorders (Cardiac disorders) | 0 (0) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/60/NCT03092960/Prot_SAP_000.pdf